CLINICAL TRIAL: NCT05231824
Title: Using Artificial Intelligence to Optimize Delivery of Weight Loss Treatment
Acronym: ReLearn
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Erica Schulte, Professor of Psychological and Brain Sciences, Drexel University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK12564
Record Dates: First submitted 2022-01-26; First posted 2022-02-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Behavioral treatment; Artificial intelligence
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BWL-S (Active Comparator): 1 year of remote gold standard, small group-based behavioral weight loss treatment with an MS-level clinician.
  Interventions: Behavioral: Standard Behavioral Weight Loss Treatment
- BWL-AI (Experimental): 1 year of remote weight loss treatment made up of a combination of (1) remote small group-based behavioral weight loss sessions, (2) 12-minute individual video calls, (2) automated text messages. An MS-level clinician will deliver the group treatment. Most video calls will be delivered by a paraprofessional coach, but some by an MS-level clinician. Each week the AI system will select one of the interventions for each participant based on which treatment the participant has responded to the best, within certain time constraints.
  Interventions: Behavioral: AI-optimized Behavioral Weight Loss Treatment

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Treatment — Behavioral weight loss treatment is the current gold standard treatment for obesity.
  Arms: BWL-S
Behavioral: AI-optimized Behavioral Weight Loss Treatment — AI-optimized Behavioral Weight Loss Treatment will continuously vary intensity (automated text message, videoconference group, individual coaching call) and coach type (paraprofessional or MS-level expert) based on continuously-monitored participant digital data.
  Arms: BWL-AI

SUMMARY:
Project ReLearn is testing the efficacy and cost-effectiveness of an Artificial Intelligence system for optimizing weight loss coaching. Participants are randomized to a 1-year weekly gold standard behavioral weight loss remote (video) group treatment or the AI-optimized treatment, which is made up of a combination of remote group treatment, short video call and automated message. In the AI-optimized condition, the system monitors outcomes (via wireless scale, mobile phone app, and wristworn tracker) and, each week, assigns each participant the treatments they have responding to the best, within certain time constraints.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be of overweight or obese BMI (27-50 kg/m)
* Individuals must be adults (aged 18-70)
* Able and willing to engage in the remote program
* Able to engage in physical activity (defined as walking two city blocks without stopping)
* Individuals must also provide consent for the research team to contact their personal physician if necessary, to provide clearance or to consult about rapid weight loss
* Access and willingness to use an Apple or Android smartphone
* Satisfactory completion of all enrollment procedures

Exclusion Criteria:

* Medical condition (e.g., cancer, type I diabetes, psychosis, full-threshold eating disorder) that may pose a risk to the participant during intervention or cause a change in weight
* Currently pregnant, breastfeeding, or planning to become pregnant in the next 12 months
* Recently began or changed the dosage of medication that can cause significant change in weight
* History of bariatric surgery
* Weight loss of > 5% in the previous 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | Baseline, 1-month, 6-month, and 12-month assessment
  Weight will be measured using the Fitbit Aria Air wireless scale, which is accurate to 0.2 kg. In order to maximize accuracy, we will (1) provide instructions (e.g., place scale on flat, hard surface; weigh upon waking, without clothes, after using the bathroom), (2) require participants to confirm that they are following instructions at each assessment point, (3) use an average of 5 consecutive daily weights for each timepoint, (4) remove errant weights (e.g., >1 kg change in 1 day).
Costs | Baseline, 1-month, 6-month, and 12-month assessment
  All time spent training counselors, participants and supervising counselors, will be tracked by the project coordinator, as will time counselors spend delivering individual and group treatment. The web portal will track counselor time on the portal, e.g., reviewing food records and texting. While the basic time commitments are pre-set by condition, several factors will vary including participant no-shows, participant drop-outs, and counselor adherence to time limits.

SECONDARY OUTCOMES:
Physical Activity | Baseline, 1-month, 6-month, and 12-month assessment
  Minutes of moderate to vigorous physical activity (MVPA) will be measured via Fitbit, a consumer-grade wrist-worn activity tracker which has superior compliance and close-to-equivalent accuracy as a research-grade accelerometer. Number of days meeting MVPA goal will be used by the AI system, with MVPA minutes as a secondary outcome.
Calorie intake | Baseline, 1-month, 6-month, and 12-month assessment
  Seven days of calorie intake as derived from the Fitbit app's food log will be used as a secondary outcome. Participants will already be tracking their consumption using the app because data are used by both the coaches (per standard treatment) and the AI system.
Acceptability as Measured by Likert Self-report Scale | 6-month and 12-month assessment
  Participants will be asked to rate satisfaction with and perceived effectiveness of the program. Counselors will rate effectiveness and ease of use.

OTHER OUTCOMES:
Self-regulation capacity | Baseline and 1-month assessment
  Self-regulation capacity will be measured directly using the Brief Self-Control Scale (which has strong retest reliability and internal consistency and predicts weight loss and dietary health).
Autonomous motivation | Baseline and 1-month assessment
  Autonomous motivation will be measured by the internally consistent and valid Treatment Self-Regulation Questionnaire.
Depressive symptoms | Baseline and 1-month assessment
  Depressive symptoms will be measured with the 20-item Center for Epidemiologic Studies Depression Scale. This self-report scale is widely used and has proven reliable across a variety of demographic groups and in both clinical and nonclinical populations.
Binge eating | Baseline and 1-month assessment
  Binge eating will be measured with the Binge Eating Module of the Eating Disorders Examination (EDE), which is a well-validated, reliable measure of eating disorder symptoms that differentiates between individuals with and without Binge Eating Disorder in

CONTACTS AND LOCATIONS:
Overall Officials: Evan M Forman, PhD, Principal Investigator — Drexel University Center for Weight, Eating and Lifestyle Science
Locations (1):
- Drexel University Center for Weight, Eating and Lifestyle Science, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry M, Taylor L, Huang Z, Chwyl C, Kerrigan S, Forman E. Automated Messaging Delivered Alongside Behavioral Treatment for Weight Loss: Qualitative Study. JMIR Form Res. 2023 Nov 6;7:e50872. doi: 10.2196/50872. PMID 37930786
- [Derived] Forman EM, Berry MP, Butryn ML, Hagerman CJ, Huang Z, Juarascio AS, LaFata EM, Ontanon S, Tilford JM, Zhang F. Using artificial intelligence to optimize delivery of weight loss treatment: Protocol for an efficacy and cost-effectiveness trial. Contemp Clin Trials. 2023 Jan;124:107029. doi: 10.1016/j.cct.2022.107029. Epub 2022 Nov 23. PMID 36435427